CLINICAL TRIAL: NCT02693834
Title: Effects of Two Different Types of Ankle Foot Orthoses on Gait Outcomes in Patients With Subacute Stroke.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18863
Record Dates: First submitted 2016-02-01; First posted 2016-02-29 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2019-11

CONDITIONS: Stroke; CVA; Hemiplegia; Hemiparesis; Foot Drop
Keywords: foot drop; Subacute stroke; AFO; gait symmetry; Gait endurance
MeSH Terms: conditions — Stroke; Hemiplegia; Paresis; Peroneal Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PLS AFO first then DA AFO (Experimental): Participants will be assigned to practice with Posterior Leaf spring AFO for a week, then they will be assigned to practice with Double adjustable AFO for another week.
  Interventions: Device: Posterior Leaf spring AFO; Device: Double adjustable AFO
- DA AFO first then PLS AFO (Experimental): Participants will be assigned to practice with Double adjustable AFO for a week, then they will be assigned to practice with Posterior Leaf spring AFO for another week
  Interventions: Device: Posterior Leaf spring AFO; Device: Double adjustable AFO

INTERVENTIONS:
Device: Posterior Leaf spring AFO — Posterior Leaf Spring AFO is an over the shelf polypropylene ankle foot orthosis to assist foot drop.
Device: Double adjustable AFO — Double adjustable AFO is a custom AFO with double action metal upright joints

SUMMARY:
PURPOSE: The purpose of this study will be to identify whether patients in the subacute stage of stroke, who demonstrate foot drop, will have better gait outcomes when using a Double Adjustable AFO, or a Posterior Leaf Spring AFO. A secondary purpose will be to determine whether one week of practice significantly changes gait outcomes with either of the AFO conditions.

INCLUSION CRITERIA: Twenty participants over the age of 18, of any gender and ethnicity, diagnosed with first time unilateral stroke, 4 - 20 weeks post-stroke onset, resulting in hemiparesis with foot drop will be recruited for this study.

EXCLUSION CRITERIA:

1. Not able to receive a double adjustable AFO through their insurance
2. Unable to follow two steps commands
3. Unable to ambulate 20 feet with or without assistive device with a minimum level of assistance of contact guard assistance.
4. Cerebellar Stroke
5. Inability to ambulate prior to stroke
6. receiving chemotherapy at the time of study

OUTCOME MEASURES:

1. Six Minute walk test
2. Gait Symmetry and Gait velocity measured with GAITRite for self paced velocity walk and fast paced velocity walk.

DATA COLLECTION:

Data will be collected three times over two weeks period.

First Visit:

Demographics, Fugl-Meyer Lower Extremity Assessment of sensorimotor function, Mini Mental State Examination 6MWT and GAITRite measurements using Both types of AFO in a random order. Afterwards participant will be given one type of AFO (randomly selected) to practice walking for a week.

Second Visit: 6MWT and GAITRite measurements using the type of AFO they were practicing with. Then the other type of AFO will be given to practice walking for a week.

Third Visit: 6MWT and GAITRite measurements using the second type of AFO that they were practicing with the week prior. Patient will be asked which type of AFO they prefer to use.

DETAILED DESCRIPTION:
Introduction: Stroke is a leading cause of death and disability in the world today. About 795,000 people are diagnosed with stroke yearly in the United States. The annual cost of stroke from medical services and disability in our nation is $ 38.6 billion dollars. Gait rehabilitation is an important aspect of neurorehabilitation with focus on attaining the most functional and symmetrical gait to prevent falls from faulty gait mechanics, and to prevent sedentary life styles and associated comorbidities. Ankle foot orthoses (AFOs) are commonly prescribed in patients with stroke to address ankle and knee instabilities and to restore a normal and safe walking pattern.The effectiveness of AFOs on various gait parameters has been reported in patients with stroke, but mostly during the chronic stages of recovery. Systematic analyses have shown that use of various types of ankle foot orthoses improve walking impairments and balance, reduce energy costs, and improve knee and ankle kinematics in people in the chronic stage of stroke recovery, greater than 6 months since the onset of stroke. It is reported that the majority of the gait improvements occur within the first 6 months following the onset of stroke. However, a limited number of studies have investigated the effects of AFOs within six months of stroke onset.

Three reported studies have investigated the effects of using an AFO compared to not using an AFO within 6 months following onset of stroke. Rao et al found that the use of an AFO significantly improved gait velocity, cadence and step length on the affected and unaffected side. Hyun et al. found that using an AFO significantly improved VO2 peak and 6 minute walk test scores . Carse et al showed significant improvement in walking velocity, average step length and cadence with use of AFO. There is only one reported study which looked at the effects of using two different types of AFOs during the subacute stage of stroke, less than 6 months following onset. Results of this study showed that gait speed and knee and ankle control were significantly higher in the Chignon AFO group compared to the polypropylene AFO group. Additionally, participants in the Chignon AFO group had significantly lower spasticity than those in the polypropylene AFO group.

In a recent case series report, investigators observed that using a custom Double Adjustable AFO during the early stages of recovery after stroke resulted in more typical muscle activation patterns, gait endurance and velocity, and near normal symmetry during gait without an assistive device or an AFO in three participants. The use of this type of AFO for gait rehabilitation following stroke in the subacute stages has not been thoroughly studied.

Statement of the Problem Patients with stroke resulting in hemiparesis and foot drop are affected by gait impairments such as poor symmetry, decreased velocity, and decreased endurance. AFOs have been shown to be an effective intervention for improving gait parameters in individuals who are in the chronic stage of stroke recovery. Although, the majority of gait improvements occur within six months of stroke, the effect of early bracing with different types of AFOs on gait outcomes has not been investigated thoroughly.

Purpose of the study:

The purpose of this study will be to identify whether patients in the subacute stage of stroke, who demonstrate foot drop, will have better gait outcomes when using a Double Adjustable AFO, or a Posterior Leaf Spring AFO. A secondary purpose will be to determine whether one week of practice significantly changes gait outcomes with either of the AFO conditions.

Research Hypotheses

The research hypotheses of this study are as follows:

1. There will be a difference in gait endurance measurements, gait symmetry measurements and gait velocity measurements at baseline when using custom Double Adjustable AFO compared to a PLS AFO in patients in subacute stage of stroke.
2. There will be a difference in gait endurance measurements, gait symmetry measurements and gait velocity measurements after one week of practice when using custom Double Adjustable AFO compared to a PLS AFO in patients in subacute stage of stroke.
3. After a week of practice, there will be a difference in gait endurance measurements, gait symmetry measurements and gait velocity measurements compared to baseline measurements, when using either custom Double Adjustable AFO or a PLS AFO in patients in subacute stage of stroke.

Participants Twenty participants over the age of 18, of any gender and ethnicity, diagnosed with first time unilateral stroke, 4 - 20 weeks post-stroke onset, resulting in hemiparesis with foot drop will be recruited. The number of participants was estimated based on previously reported studies. Hyun et al found significant differences in gait endurance measured by 6MWT when using AFO compared to using no AFO with 15 participants in a similar study. In another study by Carse et al, gait velocity and gait symmetry were found to be significantly better with 8 participants.Therefore, for our study, the potential participant number was projected as 20.

Participants will be recruited through a sample of convenience from Baylor Institute of Rehabilitation locations and through word of mouth. The physical therapists at these locations will be given a brief description of the proposed study and will be asked to screen for potential participants. Participants who meet the inclusion criteria and possess none of the exclusion criteria will be asked to volunteer for the study. Each participant will read or be read their rights as human subjects and asked to sign the informed consent approved by the Institutional Review Boards of both Baylor Health Care System and Texas Woman's University prior to enrollment in this study. A Mini Mental State Examination (MMSE) will be performed to determine whether the participant has the cognitive ability to sign the informed consent. Participants will be scheduled to do data collection on the day they receive their custom double adjustable AFO at Baylor Institute for Rehabilitation, Frisco location.

Procedures:All measurements will be obtained from each participant during three testing sessions and by only one researcher to avoid inter tester reliability issues. On the first measurement day, the primary investigator will collect demographic data including age, height, weight, leg length measurements on each side, and Fugl-Meyer Lower Extremity Assessment of sensorimotor function. Then the gait outcomes will be measured using one of the two AFO conditions in random order. The participant will select the order of AFO condition by drawing out of a hat. Randomization without replacement will be used. Once the order of AFO wearing has been determined, data will be collected in the randomly selected order. Participants will be allowed to use any type of assistive device of their choice, but the same device will be used for all conditions.

First, the 6MWT will be administered with the participant wearing the first randomized AFO. Participants will be asked to ambulate as far as possible in 6 minutes at a self-selected walking velocity through a well-lit indoor corridor. A five minute seated resting will be provided. Next, gait symmetry and gait velocity measurements will be obtained using the GAITRite system. Participants will be given a practice trial walk prior to beginning of the testing. Participants will be asked to walk at their comfortable self-selected walking velocity along the walkway. They will begin walking three meters from the start of the walkway and will stop walking two meters past the end of the walkway. The beginning and end of the walking area will be marked with red tape for visibility. The verbal instruction will be "Please walk from this red line to that red line at your comfortable speed safely". A second personnel will be walking close to the participant outside of the walkway to ensure safety. After a five minute sitting break, participant will be asked to walk as fast as they can safely. The verbal instruction will be "Please walk from this red line to that red line as fast as you can safely". The GAITRite system will be able to capture both gait symmetry and gait velocity measurements with the same walk. Three trials will be performed of the self-selected velocity walk and fast paced velocity walk. The calculated mean of the three trials will be used for data analysis. After a 10 minute seated rest break, the second AFO condition will be used and measurements will be repeated in the same order described above.

To assess the effects of practice on the gait measures, AFO's will be randomized for practice. Participants will be randomized for which AFO they will wear first. Then the participant will be provided with the selected type of AFO to practice with for the following week using a prescribed wearing schedule. At the end of the one-week practice time, the primary investigator will obtain the same measurements obtained at baseline with the participant wearing the type of AFO that was used to practice the week before. The same testing conditions and order of testing that were used at baseline will be employed. Once measurements are completed, the participant will be provided with the second type of AFO and will be asked to wear for one week using the same prescribed wearing schedule as before. Final measurements will be taken after completion of the one-week practice using the second type of AFO with the same testing conditions and orders. At the conclusion of testing each participant will be asked which AFO they will prefer to use.

Data Analysis : Descriptive statistics will be calculated for all demographic data including age, height, weight, time since onset Fugl Meyer lower extremity assessment score and AFO preference. Differences in gait endurance will be analyzed using a 2x2 repeated measures ANOVA Differences in gait symmetry, and gait velocity between the two AFO conditions and two practice conditions will be analyzed using two separate 2x2 repeated measures MANOVA. If assumption of sphericity is not met, Greenhouse-Geisser statistic will be used. An alpha level of .05 will be used to determine significance of differences, with a Bonferroni correction applied as needed to protect against Type I error.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with first time unilateral stroke
* 4 - 20 weeks post-stroke onset
* resulting in hemiparesis with foot drop

Exclusion Criteria:

* Inability to receive a double adjustable AFO through their insurance
* unable to follow two steps commands
* unable to ambulate 20 feet with or without assistive device with a minimum level of assistance of contact guard assistance
* diagnosis of cerebellar stroke
* non ambulatory prior to stroke onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-01; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priya Karakkattil, MS, Principal Investigator — Texas Woman's University
Locations (1):
- Baylor Institute for rehabilitation, Frisco, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bijleveld-Uitman M, van de Port I, Kwakkel G. Is gait speed or walking distance a better predictor for community walking after stroke? J Rehabil Med. 2013 Jun;45(6):535-40. doi: 10.2340/16501977-1147. PMID 23584080
- [Background] Bourland EL, Neville MA, Pickens ND. Loss, gain, and the reframing of perspectives in long-term stroke survivors: a dynamic experience of quality of life. Top Stroke Rehabil. 2011 Sep-Oct;18(5):437-49. doi: 10.1310/tsr1805-437. PMID 22082695
- [Background] Carse B, Bowers R, Meadows BC, Rowe P. The immediate effects of fitting and tuning solid ankle-foot orthoses in early stroke rehabilitation. Prosthet Orthot Int. 2015 Dec;39(6):454-62. doi: 10.1177/0309364614538090. Epub 2014 Jun 17. PMID 24938770
- [Background] Eng JJ, Pang MY, Ashe MC. Balance, falls, and bone health: role of exercise in reducing fracture risk after stroke. J Rehabil Res Dev. 2008;45(2):297-313. doi: 10.1682/jrrd.2007.01.0014. PMID 18566947
- [Background] de Seze MP, Bonhomme C, Daviet JC, Burguete E, Machat H, Rousseaux M, Mazaux JM. Effect of early compensation of distal motor deficiency by the Chignon ankle-foot orthosis on gait in hemiplegic patients: a randomized pilot study. Clin Rehabil. 2011 Nov;25(11):989-98. doi: 10.1177/0269215511410730. Epub 2011 Jul 12. PMID 21750010
- [Background] Everaert DG, Stein RB, Abrams GM, Dromerick AW, Francisco GE, Hafner BJ, Huskey TN, Munin MC, Nolan KJ, Kufta CV. Effect of a foot-drop stimulator and ankle-foot orthosis on walking performance after stroke: a multicenter randomized controlled trial. Neurorehabil Neural Repair. 2013 Sep;27(7):579-91. doi: 10.1177/1545968313481278. Epub 2013 Apr 4. PMID 23558080
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):188-97. doi: 10.1161/CIR.0b013e3182456d46. No abstract available. PMID 22215894
- [Background] GAITRite electronic walkway technical reference, revision L. (2013.). (No. WI-02-15).CIR Systems Inc. (GAITRite technical manual)
- [Background] Harris JE, Eng JJ, Marigold DS, Tokuno CD, Louis CL. Relationship of balance and mobility to fall incidence in people with chronic stroke. Phys Ther. 2005 Feb;85(2):150-8. PMID 15679466
- [Background] Hesse, S. (2003). Rehabilitation of gait after stroke: Evaluation, principles of therapy, novel treatment approaches, and assistive devices. Topics in Geriatric Rehabilitation, 19(2), 109-126.
- [Background] Hyun CW, Kim BR, Han EY, Kim SM. Use of an ankle-foot orthosis improves aerobic capacity in subacute hemiparetic stroke patients. PM R. 2015 Mar;7(3):264-9. doi: 10.1016/j.pmrj.2014.08.944. Epub 2014 Aug 16. PMID 25134853
- [Background] Jorgensen HS, Nakayama H, Raaschou HO, Olsen TS. Recovery of walking function in stroke patients: the Copenhagen Stroke Study. Arch Phys Med Rehabil. 1995 Jan;76(1):27-32. doi: 10.1016/s0003-9993(95)80038-7. PMID 7811170
- [Background] Kwakkel G, Kollen B, Lindeman E. Understanding the pattern of functional recovery after stroke: facts and theories. Restor Neurol Neurosci. 2004;22(3-5):281-99. PMID 15502272
- [Background] Levin MF, Kleim JA, Wolf SL. What do motor "recovery" and "compensation" mean in patients following stroke? Neurorehabil Neural Repair. 2009 May;23(4):313-9. doi: 10.1177/1545968308328727. Epub 2008 Dec 31. PMID 19118128
- [Background] Lord SE, McPherson K, McNaughton HK, Rochester L, Weatherall M. Community ambulation after stroke: how important and obtainable is it and what measures appear predictive? Arch Phys Med Rehabil. 2004 Feb;85(2):234-9. doi: 10.1016/j.apmr.2003.05.002. PMID 14966707
- [Background] McCain, K. J., Smith, P. S., & Querry, R. (2012). Ankle-foot orthosis selection to facilitate gait recovery in adults after stroke: A case series. Journal of Prosthetics and Orthotics. 24 (3), 111-121.
- [Background] Pound P, Gompertz P, Ebrahim S. A patient-centred study of the consequences of stroke. Clin Rehabil. 1998 Aug;12(4):338-47. doi: 10.1191/026921598677661555. PMID 9744669
- [Background] Rao N, Chaudhuri G, Hasso D, D'Souza K, Wening J, Carlson C, Aruin AS. Gait assessment during the initial fitting of an ankle foot orthosis in individuals with stroke. Disabil Rehabil Assist Technol. 2008 Jul;3(4):201-7. doi: 10.1080/17483100801973023. PMID 18608442
- [Background] Rosa MC, Marques A, Demain S, Metcalf CD. Fast gait speed and self-perceived balance as valid predictors and discriminators of independent community walking at 6 months post-stroke--a preliminary study. Disabil Rehabil. 2015;37(2):129-34. doi: 10.3109/09638288.2014.911969. Epub 2014 Apr 23. PMID 24754638
- [Background] Rosen E, Sunnerhagen KS, Kreuter M. Fear of falling, balance, and gait velocity in patients with stroke. Physiother Theory Pract. 2005 Apr-Jun;21(2):113-20. doi: 10.1080/09593980590922299. PMID 16392464
- [Background] Schmid AA, Rittman M. Consequences of poststroke falls: activity limitation, increased dependence, and the development of fear of falling. Am J Occup Ther. 2009 May-Jun;63(3):310-6. doi: 10.5014/ajot.63.3.310. PMID 19522139
- [Background] Simons CD, van Asseldonk EH, van der Kooij H, Geurts AC, Buurke JH. Ankle-foot orthoses in stroke: effects on functional balance, weight-bearing asymmetry and the contribution of each lower limb to balance control. Clin Biomech (Bristol). 2009 Nov;24(9):769-75. doi: 10.1016/j.clinbiomech.2009.07.006. Epub 2009 Aug 8. PMID 19665825
- [Background] Slijper A, Danielsson A, Willen C. Ambulatory Function and Perception of Confidence in Persons with Stroke with a Custom-Made Hinged versus a Standard Ankle Foot Orthosis. Rehabil Res Pract. 2012;2012:206495. doi: 10.1155/2012/206495. Epub 2012 May 17. PMID 22685664
- [Background] Tyson SF, Sadeghi-Demneh E, Nester CJ. A systematic review and meta-analysis of the effect of an ankle-foot orthosis on gait biomechanics after stroke. Clin Rehabil. 2013 Oct;27(10):879-91. doi: 10.1177/0269215513486497. Epub 2013 Jun 24. PMID 23798747
- [Background] Tyson SF, Kent RM. Effects of an ankle-foot orthosis on balance and walking after stroke: a systematic review and pooled meta-analysis. Arch Phys Med Rehabil. 2013 Jul;94(7):1377-85. doi: 10.1016/j.apmr.2012.12.025. Epub 2013 Feb 12. PMID 23416220
- [Background] Watanabe Y. Fear of falling among stroke survivors after discharge from inpatient rehabilitation. Int J Rehabil Res. 2005 Jun;28(2):149-52. doi: 10.1097/00004356-200506000-00008. PMID 15900185

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 26 participants were screened for eligibility between March 2016 and October 2017 at two outpatient clinics (Pate Rehab, Dallas and Baylor Institute for Rehabilitation, Frisco) in Dallas, Texas. Out of the 26 screened participants, 3 did not meet inclusion criteria. 23 participants consented for the study.
Pre-assignment Details: Of the 23 consented participants 2 dropped out at baseline due to fatigue. 21 people completed the baseline measurements. 11 were randomized to DA AFO first week group, PLS AFO second week(1 lost to follow up) and 10 were randomized to PLS AFO first week, and DA AFO second week. 20 participants completed both arms.
Groups:
- PLS AFO First Then DA AFO: At baseline Participants were assigned to wearing PLS AFO first for all measurements. Upon completion of baseline measurements,10 participants were randomly assigned to practice wearing the PLS AFO for the first week and the same participants were randomly assigned to the DA AFO for the second week
- DA AFO First Then PLS AFO: At baseline Participants were assigned to wearing DA AFO first for all measurements. Upon completion of baseline measurements,11 participants were randomly assigned to practice wearing the DA AFO for the first week and the same 11 participants were randomly assigned to The PLS AFO for the second week. One person was lost to follow up in this group and so only 10 completed the protocol.
Period: Baseline Measurement
Arm/Group | PLS AFO First Then DA AFO | DA AFO First Then PLS AFO
Started | 12 (10 were randomized to PLS AFO first week group (2 dropped out at baseline)) | 11 (11 participants were assigned to DA AFO first group)
Completed | 10 (10 particiapnts completed wearing PLS AFO during the first week and 10 during the second week) | 11 (10 particiapnts completed wearing DA AFO during the first week and 10 the second week (1 was lost))
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Week 1 Practice
Arm/Group | PLS AFO First Then DA AFO | DA AFO First Then PLS AFO
Started | 10 (During the first week of practice, 10 participants were assigned to PLS AFO group) | 11 (During the first week of practice, 11 participants were assigned to DAAFO group)
Completed | 10 | 11
Not Completed | 0 | 0
Period: Week 2 Practice
Arm/Group | PLS AFO First Then DA AFO | DA AFO First Then PLS AFO
Started | 10 | 11
Completed | 10 | 10
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ankle Foot Orthosis: Participants will be assigned to practice with Posterior Leaf spring AFO for a week, then they will be assigned to practice with Double adjustable AFO for another week.
  Posterior Leaf spring AFO: Posterior Leaf Spring AFO is an over the shelf polypropylene ankle foot orthosis to assist foot drop.
  Double adjustable AFO: Double adjustable AFO is a custom AFO with double action metal upright joints
Arm/Group | Ankle Foot Orthosis
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Mini Mental State exam [Mean (Standard Deviation); unit: units on a scale] — Mini Mental state Exam Score were collected (Scores on the MMSE range from 0 to 30, with scores of 25 or higher being traditionally considered normal.) For the current study the average score was 29.2 with a standard deviation of 1.0. Scores ranged from 27.0 to 30.0
  units on a scale | 29.2 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Gait Endurance
Description: 6 Minute Walk test (6MWT) to assess gait endurance using DA AFO and PLS AFO
Time Frame: at baseline
Population: 6MWT using DA AFO
Measure: Mean (Standard Deviation); unit: Meter
Groups:
- Ankle Foot Orthosis: At Baseline, all participants wore both AFOs in random order and gait endurance, gait velocity and gait symmetry were assessed and compared.
Arm/Group | Ankle Foot Orthosis
Number analyzed (Participants) | 20
Meter
  with DA AFO | 203.44 (101.19)
  With PLS AFO | 195.15 (85.83)
Statistical Analysis 1: Comparison: Ankle Foot Orthosis; In order to test the difference in gait endurance,between the two AFO conditions at baseline, a paired t-test was analyzed; Test type: Other — Paired t test; p = .293, t-test, 2 sided

2. Primary Outcome: Gait Endurance
Description: 6MWT to assess gait endurance
Time Frame: 1 week of practice with DA AFO and with PLS AFO randomly
Measure: Mean (Standard Deviation); unit: Meter
Groups:
- Ankle Foot Orthosis: Participants will be assigned to practice with Posterior Leaf spring AFO for a week, then they will be assigned to practice with Double adjustable AFO for another week. The selection of AFO was randomized. Posterior Leaf spring AFO: Posterior Leaf Spring AFO is an over the shelf polypropylene ankle foot orthosis to assist foot drop.Double adjustable AFO: Double adjustable AFO is a custom AFO with double action metal upright joints.
  10 participants wore the PLS AFO for the first week of practice and 10 participants wore the DA AFO for the first week.
Arm/Group | Ankle Foot Orthosis
Number analyzed (Participants) | 20
Meter
  With DA AFO | 255.07 (99.62)
  With PLS AFO | 235.53 (88.08)
Statistical Analysis 1: Comparison: Ankle Foot Orthosis; A repeated measures ANOVA was calculated to find the differences in gait endurance between the type of AFO and practice time; Test type: Other — Repeated measures ANOVA; p = 0.077, repeated measures ANOVA — The above value was the interaction between the type of AFO and practice time
Statistical Analysis 2: Comparison: Ankle Foot Orthosis; The main effect of type of AFO; Test type: Other — Repeated measures ANOVA; p = .046, repeated measures ANOVA — main effect of the type of AFO: F(1, 19) = 4.58, ηp2= .194
Statistical Analysis 3: Comparison: Ankle Foot Orthosis; Main effect of practice; Test type: Other — Repeated measures ANOVA; p < .001, repeated measures ANOVA — main effect of practice: F(1, 19) = 43.94, ηp2 = .698

3. Secondary Outcome: Gait Symmetry
Description: Using GAITRite for Self Selected Velocity (SSV) and Fast paced Velocity (FPV) walk Step symmetry was calculated as the ratio of affected step length over unaffected step length. Step symmetry was calculated for Self Selected Velocity (SSV) and Fast paced Velocity (FPV)
Time Frame: at baseline,1 week with DA AFO, 1 week with PLS AFO
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Ankle Foot Orthosis
Number analyzed (Participants) | 20
ratio
  DA AFO SSV Baseline | 1.16 (0.27)
  PLS AFO SSV baseline | 1.18 (0.36)
  DA AFO SSV after 1 week | 1.12 (0.19)
  PLS AFO SSV after 1 week | 1.10 (0.24)
  DA AFO FPV Baseline | 1.18 (0.29)
  PLS AFO FPV Baseline | 1.22 (0.37)
  DA AFO FPV after 1 week | 1.16 (0.23)
  PLS AFO FPV after 1 week | 1.11 (0.23)
Statistical Analysis 1: Comparison: Ankle Foot Orthosis; The significance of differences in gait symmetry, between the two AFO conditions at baseline were analyzed using a paired t test for self selected velocity; Test type: Other — paired t test; p = .688, t-test, 2 sided
Statistical Analysis 2: Comparison: Ankle Foot Orthosis; The significance of differences in gait symmetry at self select velocity, between the two AFO conditions and two practice conditions were analyzed using repeated measures MANOVA; Test type: Other — repeated measures MANOVA; p = .397, repeated measures MANOVA — The above p value is for the interaction effects between type of AFO and practice time for gait symmetry at the self selected velocity F(1, 19)= 0.75, ηp2 = .038
Statistical Analysis 3: Comparison: Ankle Foot Orthosis; Main effect of AFO on gait symmetry was analyzed at self selected velocity; Test type: Other — A repeated measures MANOVA; p = .950, Repeated measures MANOVA — Main effect of AFO on gait symmetry at SSV: F(1, 19) = 0.004, ηp2 =.00
Statistical Analysis 4: Comparison: Ankle Foot Orthosis; Main effect of practice on gait symmetry at Self selected velocity; Test type: Other — Repeated measures MANOVA; p = .111, repeated measures MANOVA — The main effect of practice on gait symmetry at self selected velocity F(1, 19) = 2.79, ηp2 = .128
Statistical Analysis 5: Comparison: Ankle Foot Orthosis; The significance of differences in gait symmetry, between the two AFO conditions at baseline were analyzed using a paired t test for fast paced velocity; Test type: Other; p = .260, t-test, 2 sided
Statistical Analysis 6: Comparison: Ankle Foot Orthosis; The significance of differences in gait symmetry at fast paced velocity, between the two AFO conditions and two practice conditions were analyzed using repeated measures MANOVA; Test type: Other — repeated measures MANOVA; p = .113, repeated measures MANOVA — The above p value is for the interaction effects between type of AFO and practice time for gait symmetry at fast paced velocity FPV F(1, 19) = 2.76,, ηp2 = .127
Statistical Analysis 7: Comparison: Ankle Foot Orthosis; The main effect of AFO on gait symmetry at fast paced velocity walk was assessed with repeated measures MANOVA; Test type: Other — Repeated measures MANOVA; p = .918, repeated measures MANOVA — The main effect of AFO on gait symmetry at fast paced velocity: F(1, 19) = 0.01, ηp2 = 0.001
Statistical Analysis 8: Comparison: Ankle Foot Orthosis; The main effect of practice on gait symmetry at fast paced velocity walk was assessed with repeated measures MANOVA; Test type: Other — Repeated measures MANOVA; p = .077, repeated measures MANOVA — The main effect of practice on gait symmetry at fast paced velocity: F(1, 19) = 3.50, ηp2 = .155

4. Secondary Outcome: Gait Velocity SSV and FPV
Description: using GAITRite for Self selected velocity (SSV)walk and fast paced velocity (FPV) walk
Time Frame: at baseline,1 week with DA AFO, 1 week with PLS AFO
Measure: Mean (Standard Deviation); unit: meter per sec
Arm/Group | Ankle Foot Orthosis
Number analyzed (Participants) | 20
meter per sec
  DA AFO SSV Baseline | 0.58 (0.26)
  PLS AFO SSV baseline | 0.58 (0.26)
  DA AFO SSV after 1 week | 0.70 (0.29)
  PLS AFO SSV after 1 week | 0.66 (0.27)
  DA AFO FPV Baseline | 0.80 (0.38)
  PLS AFO FPV Baseline | 0.78 (0.36)
  DA AFO FPV after 1 week | 0.95 (0.36)
  PLS AFO FPV after 1 week | 0.91 (0.35)
Statistical Analysis 1: Comparison: Ankle Foot Orthosis; The significance of differences in gait velocity at self select velocity, between the two AFO conditions and two practice conditions were analyzed using repeated measures MANOVA; Test type: Other — A repeated measures MANOVA; p = .209, Repeated measures MANOVA — The above p value is for the interaction effects between the type of AFO and practice time at self selected velocity: F(1, 19) = 1.69, ηp2 = .082
Statistical Analysis 2: Comparison: Ankle Foot Orthosis; Main effect of AFO on gait velocity was analyzed at self selected velocity; Test type: Other — Repeated measures MANOVA; p = .32, repeated measures MANOVA — Main effect of AFO on gait velocity at self selected velocity: F(1, 19) = 1.05, ηp2 = .05
Statistical Analysis 3: Comparison: Ankle Foot Orthosis; Main effect of Practice on gait velocity was analyzed at self selected velocity; Test type: Other — Repeated measures MANOVA; p = .001, repeated measures MANOVA — Main effect of practice on gait velocity at self selected velocity:F(1, 19) = 14.38, ηp2 = .431
Statistical Analysis 4: Comparison: Ankle Foot Orthosis; The significance of differences in gait velocity at fast paced velocity, between the two AFO conditions and two practice conditions were analyzed using repeated measures MANOVA; Test type: Other — repeated measures MANOVA; p = .280, repeated measures MANOVA — The above p value is for the interaction effects between the type of AFO and practice time at fast paced velocity: F( 1, 19) = 1.24, ηp2 = .61
Statistical Analysis 5: Comparison: Ankle Foot Orthosis; Main effect of AFO on gait velocity was analyzed for self selected velocity; Test type: Other — repeated measures MANOVA; p = .072, repeated measures MANOVA — Main effect of AFO on gait velocity was analyzed at self selected velocity:FPV F(1, 19) = 3.63, ηp2 =.16
Statistical Analysis 6: Comparison: Ankle Foot Orthosis; Main effect of Practice on gait velocity was analyzed for fast paced velocity; Test type: Other — Repeated measures MANOVA; p < .001, repeated measures MANOVA — Main effect of Practice on gait velocity for fast paced velocity: F(1, 19) = 23.73, ηp2 = .555

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the entire study enrollment time, for 3 weeks.
Description: One participant could not complete baseline assessment due to fatigue associated with chemotherapy. IRB was contacted and a new exclusion criteria was added to exclude participants who were currently undergoing chemotherapy at the time of data collection.
  One participant had another stroke while at home before the final measurement during the second week of practice with the PLS AFO. This was not related to the study intervention, IRB was informed
Groups:
- PLS AFO: Posterior Leaf Spring AFO
- DA AFO: Double Adjustable AFO
Arm/Group | PLS AFO | DA AFO
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/23
Other Adverse Events (participants affected / at risk) | 1/23 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLS AFO (N=23) | DA AFO (N=23)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) — One participant had another stroke while at home before the final measurement. This event was unrelated to the intervention used.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLS AFO (N=23) | DA AFO (N=23)
Fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — one participant got fatigued and could not continue testing on first day due to side effect of chemo

LIMITATIONS AND CAVEATS:
Limited sample size Use of repeated measures design

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT02693834/Prot_SAP_000.pdf